CLINICAL TRIAL: NCT03665636
Title: Anaplerotic Therapy Using Triheptanoin for Patients With Glycogen Storage Disease Type I
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Areeg El-Gharbawy (Other)
Collaborators: Ultragenyx Pharmaceutical Inc (Industry)
Responsible Party: Sponsor-Investigator, Areeg El-Gharbawy, Assistant Professor of Pediatrics, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00103582
Record Dates: First submitted 2018-08-23; First posted 2018-09-11 (Actual); Last update posted 2021-12-15 (Actual); Status verified 2021-12

CONDITIONS: Glycogen Storage Disease Type I
Keywords: Glycogen Storage Disease Type I; GSD I; Anaplerosis; Triheptanoin; Hypoglycemia
MeSH Terms: conditions — Glycogen Storage Disease Type I; Hypoglycemia | interventions — triheptanoin

STUDY DESIGN:
Intervention Model Description: This study is an interventional, open-label, feasibility pilot project to study the safety, efficacy, and tolerability of triheptanoin in patients with GSD I.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Triheptanoin (Experimental): Open Label Study
  Interventions: Drug: Triheptanoin

INTERVENTIONS:
Drug: Triheptanoin — This is an open-label study. The UX007 (triheptanoin) starting dose will be 0.25 - 0.5 g/kg and titrated to a maximum of 2.5g/kg depending the on the subject's tolerance. The dose may be reduced if not tolerated. The compound will be administered 3-4 times per day, either at the end of a meal or with a snack. It should be given at least 2 hours apart from any cornstarch dose to allow each to act independent of one another, and to prevent the risk of increased gastrointestinal side effects. The doses may be held during episodes of gastroenteritis or diarrhea.
  Other Names: UX007

SUMMARY:
This study will be an open-label, prospective, interventional feasibility pilot project to study the efficacy, safety, and tolerability of UX007 (triheptanoin) on reducing hypoglycemic events in patients with GSD I. Subjects will serve as their own control. Five (5) subjects who are treatment naïve to UX007 (triheptanoin) and are already on standard dietary therapy for GSDI will be enrolled.

The primary objective is to evaluate the efficacy, safety, and tolerability of UX007 (triheptanoin) in patients with GSD I. The secondary objectives include evaluating the effect of UX007 (triheptanoin) on maintaining the duration of normoglycemia between meals based on glucose monitoring (Preventing and reducing the frequency of hypoglycemia); reduction/stabilization of the dose of cornstarch; and the prevention of increased liver steatosis based on ultrasound with elastography.

DETAILED DESCRIPTION:
Prior to first study appointment:

A medical record review will be done prior to the appointment to confirm the diagnosis of GSD I. For interested subjects who are not already known to the investigators (i.e., patients of the Duke University Medical Center), a release of protected health information will be signed by the potential subjects to obtain records that can be used to confirm diagnosis.

Baseline / Visit 1:

Study subjects will be instructed to come to the DUMC to review and sign the informed consent document. At that time, complete medical history and complete physical examination will be obtained. Blood and urine will be collected for laboratory assessments. Height, weight, and vital signs (blood pressure, pulse, respiration) will be collected.

A nutritional history and review of diet dairy collected three days prior to the visit will be reviewed by a study dietitian. The blood glucose monitoring log for the three days prior to the visit will also be reviewed the study dietitian and MD. Study staff will collect concomitant medications and adverse event collection will begin once dosing with UX007 is initiated. An ultrasound with elastography will be conducted at the DUMCs radiology department and reviewed and a report generated by a radiologist.

Safety Phone Contact:

Subjects will be called by study staff the day after they start the UX007 and again 4 weeks later to assess nutritional history, review of glucose diary, review of dosing compliance, and to obtain an updated weight. Study staff will also review adverse events (AE/SAE) and concomitant medications during these calls. If a subject experiences an AE/SAE they will be contacted every two weeks until the AE/SAE is resolved.

2, 4, and 6 Month/Early Termination Visits:

Same procedures will be conducted as at the baseline visit, with the exception of the ultrasound with elastography, which will only be collected again at the 6 Month/Early Termination Visit.

Post-termination Phone Contact:

2-6 weeks after the 6 month/early termination visit study staff will contact the subject to collect an interim medical history, evaluation of nutritional history, review of glucose diary as well as review of adverse events and concomitant medications. An updated weight will also be obtained.

ELIGIBILITY:
Inclusion Criteria:

* Naive to UX007 (triheptanoin)
* Confirmed documented diagnosis of GSDI: confirmation may be based on mutation analysis, liver biopsy, or enzyme testing
* Willing and able to complete all aspects of the study through the end of the study, including visits and tests, documentation of symptoms, blood sugar and dietary log, and administration of UX007 (triheptanoin); minors in the study must have a parent/legally authorized representative who is willing and able to assist in all applicable study requirements

Exclusion Criteria:

* Have a history of severe inflammatory bowel disease, or severe chronic diarrhea per the PI discretion on conventional doses of cornstarch
* Patient is on any other form of medium chain triglyceride (MCT) during the time of the study. Patients will be asked to stop any nutritional compound that includes MCT oil one week (7 days) prior to baseline.
* Have any co-morbid conditions, including major organ-system disease(s) that in the opinion of the Investigator, places the subject at increased risk of complications, interferes with study participation or compliance, or confounds study objectives
* Pregnancy
* Patients on continuous feeds, with a diagnosis of diabetes, and/or a diagnosis of any other inborn error or metabolism

Ages: 1 Month to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2020-10-16 (Actual); Primary Completion 2021-10-21 (Actual); Study Completion 2021-10-21 (Actual)

PRIMARY OUTCOMES:
Blood glucose level | Baseline and 6 months
  Reviewing the change in blood glucose levels from baseline to 6 month visit

SECONDARY OUTCOMES:
Dietary intake | Baseline and 6 months
  Reviewing the change in fat, protein, and carbohydrate intake, after adding the intervention, from baseline to 6 month visit
Liver steatosis assessment | Baseline and 6 months
  Reviewing the change fatty infiltration (steatosis) using ultrasound elastography from baseline to 6 months visit. This technique will the degree of steatosis which is reflected by echogenicity and stiffness that is measured by 2D ultrasound shear wave speed measurements.
Liver size assessment | Baseline and 6 months
  Reviewing the change in liver size using ultrasound elastography from baseline to 6 months visit. This technique will provide liver size at both timepoints.
Laboratory metabolic control markers | Baseline and 6 months
  Reviewing laboratory markers indicative of metabolic control which include glucose, triglycerides, and uric acid measured in mg/dl from baseline to 6 month visit
Other laboratory metabolic control markers | Baseline and 6 months
  Reviewing lactate levels as a main indicator of metabolic control measured in mMol/L from baseline to 6 month visit

CONTACTS AND LOCATIONS:
Overall Officials: Areeg El-Gharbawy, MD, Principal Investigator — Duke University, Department of Pediatrics - Medical Genetics
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chou JY, Matern D, Mansfield BC, Chen YT. Type I glycogen storage diseases: disorders of the glucose-6-phosphatase complex. Curr Mol Med. 2002 Mar;2(2):121-43. doi: 10.2174/1566524024605798. PMID 11949931
- [Background] Fernandes J, Pikaar NA. Ketosis in hepatic glycogenosis. Arch Dis Child. 1972 Feb;47(251):41-6. doi: 10.1136/adc.47.251.41. PMID 4336232
- [Background] Rasmussen BB, Holmback UC, Volpi E, Morio-Liondore B, Paddon-Jones D, Wolfe RR. Malonyl coenzyme A and the regulation of functional carnitine palmitoyltransferase-1 activity and fat oxidation in human skeletal muscle. J Clin Invest. 2002 Dec;110(11):1687-93. doi: 10.1172/JCI15715. PMID 12464674
- [Background] Das AM, Lucke T, Meyer U, Hartmann H, Illsinger S. Glycogen storage disease type 1: impact of medium-chain triglycerides on metabolic control and growth. Ann Nutr Metab. 2010;56(3):225-32. doi: 10.1159/000283242. Epub 2010 Mar 30. PMID 20357432
- [Background] Nagasaka H, Hirano K, Ohtake A, Miida T, Takatani T, Murayama K, Yorifuji T, Kobayashi K, Kanazawa M, Ogawa A, Takayanagi M. Improvements of hypertriglyceridemia and hyperlacticemia in Japanese children with glycogen storage disease type Ia by medium-chain triglyceride milk. Eur J Pediatr. 2007 Oct;166(10):1009-16. doi: 10.1007/s00431-006-0372-0. Epub 2007 Jan 6. PMID 17206455
- [Background] Gu L, Zhang GF, Kombu RS, Allen F, Kutz G, Brewer WU, Roe CR, Brunengraber H. Parenteral and enteral metabolism of anaplerotic triheptanoin in normal rats. II. Effects on lipolysis, glucose production, and liver acyl-CoA profile. Am J Physiol Endocrinol Metab. 2010 Feb;298(2):E362-71. doi: 10.1152/ajpendo.00384.2009. Epub 2009 Nov 10. PMID 19903863
- [Background] Farah BL, Sinha RA, Wu Y, Singh BK, Lim A, Hirayama M, Landau DJ, Bay BH, Koeberl DD, Yen PM. Hepatic mitochondrial dysfunction is a feature of Glycogen Storage Disease Type Ia (GSDIa). Sci Rep. 2017 Mar 20;7:44408. doi: 10.1038/srep44408. PMID 28317891
- [Background] Roe CR, Mochel F. Anaplerotic diet therapy in inherited metabolic disease: therapeutic potential. J Inherit Metab Dis. 2006 Apr-Jun;29(2-3):332-40. doi: 10.1007/s10545-006-0290-3. PMID 16763896